CLINICAL TRIAL: NCT00046254
Title: Evaluating the Ability of Zoledronic Acid to Reduce the Rate of Subsequent Osteoporotic Fractures After a Hip Fracture
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CZOL446H2310
Record Dates: First submitted 2002-09-24; First posted 2002-09-25 (Estimated); Last update posted 2012-05-02 (Estimated); Status verified 2012-05

CONDITIONS: Osteoporosis; Hip Fracture
Keywords: hip fracture; recurrent fracture; fracture; bone loss; bisphosphonate; bone mineral density; osteoporosis; zoledronic acid; geriatrics; rehabilitation; elderly; nursing home; orthopedic
MeSH Terms: conditions — Osteoporosis; Hip Fractures; Fractures, Bone; Bone Diseases, Metabolic | interventions — Zoledronic Acid

INTERVENTIONS:
Drug: Zoledronic Acid

SUMMARY:
The purpose of this study is to evaluate whether zoledronic acid given once yearly for two years to men and women after surgical repair of a recent hip fracture will significantly reduce the rate of all re-occurring (new) osteoporotic fractures. All patients will receive vitamin D and calcium.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ages 50 years or older
* Must have a recent hip fracture repair in the past 90 days
* Must be able to walk with or without assistive device (for example, using a walker) prior to the hip fracture

Exclusion Criteria:

* Current bisphosphonate users such as aredia (pamidronate), didronel (etidronate), fosamax (alendronate), actonel (residronate), skelid (tiludronate)

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2127
Dates: Start 2002-02; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Significant reduction in rate of clinical fractures after surgical repair of hip fracture

SECONDARY OUTCOMES:
Increase in total hip and femoral neck BMDs

CONTACTS AND LOCATIONS:
Locations (28):
- United States (27):
  - University of Alabama Hospital, Birmingham, Alabama
  - Osteoporosis Diagnostic Center, Eureka, California
  - Sharp Grossmont Hosptial, La Mesa, California
  - The Permanente Group, Santa Rosa, California
  - Radiant Research Lake Worth, Lake Worth, Florida
  - Atlanta Resarch Center, Decatur, Georgia
  - United Osteoporosis Center Health Services, Gainesville, Georgia
  - Galesburg Orthopedic Services LTD, Galesburg, Illinois
  - Illinois Bone and Joint Institute, Morton Grove, Illinois
  - Mercy Arthritis and Osteoporosis Center, Des Moines, Iowa
  - Maine Medical Center Research Institute, Portland, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Wayne State University, Div. of Endocrinology, Detroit, Michigan
  - Health East Osteoporosis Service, Woodbury, Minnesota
  - Highland Hospital, Rochester, New York
  - University of North Carolina Hospital, Chapel Hill, North Carolina
  - Duke University Health System, Durham, North Carolina
  - University Orthopaedics, Canfield, Ohio
  - Ohio State University, Columbus, Ohio
  - University of Pennsylvania Health System-Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Saint Joseph Medical Center, West Reading, Pennsylvania
  - Saint Josephs, Warwick, Rhode Island
  - Palmetto Richland Memorial Hospital, Columbia, South Carolina
  - Seton Medical Center, Austin, Texas
  - St. Luke's Episcopal Hospital, Houston, Texas
  - Danville Regional Medical Center, Danville, Virginia
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
- Novartis, Nuremberg, Germany

REFERENCES:
- [Derived] Magaziner JS, Orwig DL, Lyles KW, Nordsletten L, Boonen S, Adachi JD, Recknor C, Colon-Emeric CS, Mesenbrink P, Bucci-Rechtweg C, Su G, Johnson R, Pieper CF. Subgroup variations in bone mineral density response to zoledronic acid after hip fracture. J Bone Miner Res. 2014 Dec;29(12):2545-51. doi: 10.1002/jbmr.2283. PMID 24839241
- [Derived] Prieto-Alhambra D, Judge A, Arden NK, Cooper C, Lyles KW, Javaid MK. Fracture prevention in patients with cognitive impairment presenting with a hip fracture: secondary analysis of data from the HORIZON Recurrent Fracture Trial. Osteoporos Int. 2014 Jan;25(1):77-83. doi: 10.1007/s00198-013-2420-8. Epub 2013 Jun 28. PMID 23812596
- [Derived] Adachi JD, Lyles KW, Colon-Emeric CS, Boonen S, Pieper CF, Mautalen C, Hyldstrup L, Recknor C, Nordsletten L, Moore KA, Bucci-Rechtweg C, Su G, Eriksen EF, Magaziner JS. Zoledronic acid results in better health-related quality of life following hip fracture: the HORIZON-Recurrent Fracture Trial. Osteoporos Int. 2011 Sep;22(9):2539-49. doi: 10.1007/s00198-010-1514-9. Epub 2011 Jan 20. PMID 21249332
- [Derived] Grbic JT, Black DM, Lyles KW, Reid DM, Orwoll E, McClung M, Bucci-Rechtweg C, Su G. The incidence of osteonecrosis of the jaw in patients receiving 5 milligrams of zoledronic acid: data from the health outcomes and reduced incidence with zoledronic acid once yearly clinical trials program. J Am Dent Assoc. 2010 Nov;141(11):1365-70. doi: 10.14219/jada.archive.2010.0082. PMID 21037195
- [Derived] Lyles KW, Colon-Emeric CS, Magaziner JS, Adachi JD, Pieper CF, Mautalen C, Hyldstrup L, Recknor C, Nordsletten L, Moore KA, Lavecchia C, Zhang J, Mesenbrink P, Hodgson PK, Abrams K, Orloff JJ, Horowitz Z, Eriksen EF, Boonen S; HORIZON Recurrent Fracture Trial. Zoledronic acid and clinical fractures and mortality after hip fracture. N Engl J Med. 2007 Nov 1;357(18):1799-809. doi: 10.1056/NEJMoa074941. Epub 2007 Sep 17. PMID 17878149